CLINICAL TRIAL: NCT04179448
Title: A Prospective, Randomized Clinical Trial to Compare Side Access Mucosal Releasing Incision (SAMRI) and Sulcular Tunnel Access Procedures With Coronally Advanced Flap and Acellular Dermal Matrix (ADM) to Treat Gingival Recession.
Brief Title: A Comparison of Side Access Mucosal Releasing Incision (SAMRI) and Sulcular Tunnel Access to Treat Gingival Recession.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria L. Geisinger, DDS, MS, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAMRI IRB-300004045; UAB-Perio (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gingival Recession; Lack of Keratinized Gingiva
Keywords: Keratinized Tissue; Keratinized Gingiva; Gingival recession; Mucogingival defect; SAMRI; Acellular Dermal Matrix; Sulcular tunnel technique; Patient-centered outcomes
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Side Access Mucosal Releasing Incision (SAMRI) (Experimental): SAMRI incision to allow for coronally advanced flap and placement of acellular dermal matrix (ADM) graft
  Interventions: Procedure: SAMRI
- Sulcular Tunnell access (Active Comparator): Sulcular tunnel access incision to allow for coronally advanced flap and placement of acellular dermal matrix (ADM) graft
  Interventions: Procedure: STA

INTERVENTIONS:
Procedure: SAMRI — Side Access Mucosal Releasing Incision (SAMRI) will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
  Arms: Side Access Mucosal Releasing Incision (SAMRI)
Procedure: STA — Sulcular tunnel access incision will be performed on all individuals in this arm of the study to facilitate coronal advancement of the gingival flap and placement of acellular dermal matrix
  Arms: Sulcular Tunnell access

SUMMARY:
This study will compare two incision designs to allow for coronal gingival/mucosal flap advancement and tissue augmentation with acellular dermal matrix (ADM) graft around teeth with gingival recession and a lack of adequate keratinized gingiva.

The SAMRI technique described is a novel technique involving a simplified incision and suturing technique and to the investigators' knowledge, this is the first study that seeks to compare this technique to other techniques for differences in clinical outcomes (percentage root coverage, resultant tissue thickness, and width of keratinized tissue) and patient-centered outcomes (post-operative pain, swelling, changes in daily activities, and patient-assessed esthetics) in a controlled study.

DETAILED DESCRIPTION:
Research data and daily clinical observations reveal that teeth with gingival recession and a lack of adequate keratinized tissue (KT) are more prone to persistent gingival inflammation, dentinal sensitivity, radicular (root) caries (tooth decay), faster periodontal attachment loss, and compromised plaque control. Soft tissue grating (by various techniques) aims at changing the quality, quantity and placement of the soft tissue around teeth by covering exposed root surfaces and creating or increasing the zone of keratinized mucosa (KM) surrounding the affected teeth. Both techniques tested have shown good clinical outcomes with regard to root coverage, but clinical reports suggest that decreased intrasurgical time and the simplified protocol of the SAMRI technique may result in improved clinical outcomes and/or a decrease in postoperative morbidity and complications as assessed by patients.

Specific aims for this project include the evaluation of:

* Percentage of root coverage at 6 and 12 months following grafting with SAMRI and sulcular tunnel access with ADM
* KT width at 6 and 12 month following grafting with SAMRI and sulcular tunnel access with ADM
* Change in tissue thickness of the grafted sites at 6 and 12 months
* Practitioner-assessed esthetic outcomes using a standardized pink esthetic scale (PES) at 6 and 12 months postoperatively
* Patient-assessed esthetic outcomes at 6 and 12 months post-operatively
* Patient centered outcomes including pain, bleeding, swelling, change in daily activities at 1 week and 1 month postoperatively

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* At least 18 years old
* Must be a patient of the UAB Dental School
* Able to read and understand informed consent document
* One or more adjacent teeth (up to four) with Miller class I or II gingival recession defects and less than or equal to 2mm of KT at each site to be treated.
* Presence of periodontally healthy, non-carious neighboring teeth, healthy implants or edentulous ridges on either side of the involved site(s)
* No anticipated need for restorative care at the teeth to be treated during the study period.

Exclusion Criteria:

* Non-English speaking
* Less than 18 years old
* Smokers/tobacco users (>10 cigarettes/day)
* Patients with systemic pathologies or conditions contraindicating oral surgical procedures or adversely affecting wound healing
* Presence of active periodontal disease or radiographic interproximal bone loss or tooth malposition, which would yield a Miller class III or IV categorization for the recession defect.
* Presence of frenulae or other soft tissue anomalies at the site(s) to be treated that, in the opinion of the investigators, will interfere with successful access and treatment of the soft tissue defects.
* Previous soft tissue grafting at the site(s) to be treated

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of root coverage at 6 and 12 months following grafting with SAMRI and sulcular tunnel access with ADM | From baseline to 6 months and 12 months
  Compare the change in the exposed root surface at sites with gingival recession.

SECONDARY OUTCOMES:
KT width at 6 and 12 month following grafting with SAMRI and sulcular tunnel access with ADM | From baseline to 6 and 12 months
  Compare the change in keratinized tissue (KT) between two incision designs for root coverage and tissue augmentation.
Change in tissue thickness of the grafted sites at 6 and 12 months | From baseline to 6 and 12 months
  Using a periodontal probe, soft tissue thickness will be measured (in mm) and compared between FGG and CTG following soft tissue grafting.
Assessed esthetic outcomes using a standardized pink esthetic scale (PES) at 6 and 12 months postoperatively | From baseline to 6 and 12 months
  Assess esthetic outcomes using an established periodontal esthetic score (PES). This score evaluates the color of the gum utilizing 5 subscales ranging from 0(worse) to 2 (better) allowing for a summed total score of 10.
Assessed esthetic outcomes at 6 and 12 months post-operatively | At 6 and 12 months postoperatively
  A visual analogue scale (VAS) based questionnaire regarding esthetic appearance, pain, swelling, bruising, effects on daily activities will be administered. This measurement ranges from 0-10 (0 being better and 10 being worse).
Patient centered outcomes including pain, bleeding, swelling, change in daily activities at 1 week and 1 month postoperatively | 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months postoperatively.
  A visual analogue scale (VAS) based questionnaire regarding esthetic appearance, pain, swelling, bruising, effects on daily activities. This measurement ranges from 0-10 (0 being better and 10 being worse).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Geisinger, DDS, MS, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be shared with other researchers outside of our research laboratory group.